CLINICAL TRIAL: NCT07330752
Title: PRemarket INvestigation to Evaluate the Clinical Safety and effectIveness of the Protective "A3- Shield" System for the stabIlIzation of Abdominal Aortic aneurysmS - Pilot Phase
Brief Title: First-in-Human Trial of the A3-Shield System for Stabilizing Abdominal Aortic Aneurysms
Acronym: PRINCIPIIS-FIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Angiolutions GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-P001-2025
Record Dates: First submitted 2025-11-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Aneurysm, Abdominal Aortic
Keywords: A3-Shield; Small AAA; Pulse Wave Modulation
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device implantation (Experimental): A3-Shield Implantation
  Interventions: Device: A3-Shield Implantation

INTERVENTIONS:
Device: A3-Shield Implantation — Implantation of the A3-Shield Device in the AAA Neck

SUMMARY:
This clinical trial evaluates the safety and feasibility of the A3-Shield implant for stabilising small abdominal aortic aneurysms in adult patients. The study enrolls men and women with small, asymptomatic infrarenal abdominal aortic aneurysms who are eligible for an elective catheter-based procedure.

The trial aims to determine whether implantation of the A3-Shield device is technically feasible and whether it is associated with mechanical immobilization of the aneurysm neck. The study also assesses the peri-procedural and safety profile of the device.

Participants will undergo implantation of the A3-Shield device and attend scheduled follow-up visits that include clinical assessments and imaging such as ultrasound and computed tomography. The study does not include randomisation or a separate control group.

DETAILED DESCRIPTION:
Current management of abdominal aortic aneurysms is severely limited by the lack of therapeutic options that can halt the underlying dilating biology. At present, there is no available intervention that can sufficiently intercept the size progression of small abdominal aortic aneurysms. This gap is highly relevant because the vast majority of abdominal aortic aneurysms are detected at a small size, and a substantial proportion of these aneurysms enlarge over the following years and eventually require prosthetic repair, which carries procedure-related and long-term risks. The limited efficacy of endovascular aortic repair in small aneurysms and the significant long-term complications observed in large aneurysms treated by endovascular aortic repair are thought to be related, at least in part, to insufficient control of aneurysm sac expansion. Effective stabilisation of aneurysm size at an early stage therefore represents a major unmet need in abdominal aortic aneurysm management.

The A3-Shield implant introduces a new approach to aneurysm treatment by targeting the biomechanical forces that contribute to aneurysm enlargement. Each heartbeat generates aortic pulse waves that propagate along the vessel and induce pulsatile wall motion. As these pulse waves reach the aneurysmal segment, they generate concentrated mechanical stress at the AAA shoulder region. This stress concentration is believed to promote further expansion of the aneurysm. The A3-Shield implant is designed to counteract this mechanism by mechanically immobilizing the aneurysm neck and gradually dampening the transmission of harmful pulse wave forces into the aneurysm sac, thereby aiming to protect the aneurysm from stress-induced enlargement.

This first-in-human clinical trial evaluates the safety and feasibility of the A3-Shield implant in adult patients with small infrarenal abdominal aortic aneurysms. The primary objectives are to determine whether the implantation procedure is technically feasible and whether it is associated with suppression of pulse wave transmission at the aneurysm neck. The study also assesses the peri-procedural and safety profile of the device.

Participants undergo a catheter-based implantation of the A3-Shield device under fluoroscopic guidance. Following the procedure, they attend scheduled follow-up visits that include clinical examinations and imaging such as ultrasound and computed tomography. The study does not include randomisation or a separate control group.

The findings from this pilot phase are intended to support further clinical development and may provide early evidence for a new interventional strategy that addresses an unmet need in the management of small abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

IC1. Male and female subjects ≥ 18 years at the time of screening. Female subjects must be of non-childbearing potential or otherwise not pregnant and not planning to become pregnant during the study follow-up period.

IC2. Subject has a documented fusiform infrarenal abdominal aortic aneurysm characterized by the following:

* Aneurysm size of 3.0-5.0 cm in maximum diameter for males; 3.0 - 4.5 for females (diameter measured in CTA perpendicular to the line of flow)
* Aortic neck diameter ≥17mm and ≤ 29mm
* Adequate landing zone for a tubular device of ≥ 30 mm length

IC3. Access vessel size and morphology allows endovascular access of 14F (or larger) introducer sheaths and catheters

IC4. Subject (or legal representative) understands the study requirements and the procedures and provided written informed consent.

IC5. Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow-up visits.

Exclusion Criteria:

EC1. Subject has an aneurysm that is:

* symptomatic
* ruptured
* thoracic
* suprarenal
* thoraco-abdominal
* isolated ilio-femoral
* mycotic
* inflammatory
* pseudoaneurysmatic
* traumatic

EC2. Subject has any type of aortic dissection.

EC3. Subject has congenital connective tissue disease, e.g., Marfan's Syndrome or Ehlers-Danlos Syndrome.

EC4. Subject has significant (>25% of vessel circumference of aortic neck) aortic mural thrombus at the attachment site that could compromise fixation of the device.

EC5. Subject has arterial access that is not acceptable for the device delivery systems as defined in the device Instructions For Use.

EC6. Subject has had an acute myocardial infarction within 180 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin elevation).

EC7. Subject has untreated coronary artery disease, which in the opinion of the treating physician, is clinically significant and requires revascularization.

EC8. Subject has congestive heart failure (NYHA class III or IV) or high-grade valvular disease.

EC9. Subject has had a cerebrovascular accident or transient ischemic attack within the past 90 days prior to study enrollment.

EC10. Subject has end-stage renal disease or has a creatinine > 2.0 mg/dl or is on dialysis.

EC11. Subject has a history of bleeding diathesis or coagulopathy.

EC12. Subject has Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.

EC13. Subject has had or plans to have an unrelated major surgical or interventional procedure (including trans-aortic interventions) within 30 days prior or post implantation of the device.

EC14. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated or has known hypersensitivity to the device components.

EC15. Subject is participating in another investigational drug or device study and has not completed the follow-up required for that study at least 30 days prior to signing the informed consent form in this study.

EC16. Subject is morbidly obese (body mass index ≥ 40 kg/m2) or has other documented conditions that inhibit radiographic visualization of the aorta.

EC17. Subject has an active infection or chronic systemic illness at the time of the index procedure that may interfere with study objectives.

EC18. Subject has current problems with substance abuse.Smoking is NOT an exclusion criterion.

EC19. Subject has severe incapacitating dementia.

EC20. Subject has a life expectancy of less than 24 months due to comorbid conditions based on the assessment of the investigator at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint: Absence of Major Adverse Events | Within 30 days of the index procedure
  Absence of Major Adverse Events (MAEs). MAE is defined as a composite of death, stroke, myocardial infarction, new onset renal failure (requiring dialysis), respiratory failure (requiring mechanical ventilation), paralysis or paraparesis, bowel ischemia requiring surgical intervention or procedural blood loss ≥ 1,000 cc.
Primary effectiveness endpoint: Successful aneurysm treatment | Conclusion of the index procedure
  Successful aneurysm treatment defined as the composite of
  1. Technical success, defined as successful insertion of the delivery system through the vasculature, successful deployment of the device at the intended location, and successful removal of the delivery system
  2. Immobilization of the distal AAA neck, defined as aortic circumferential cyclic strain < 10% as measured via vascular ultrasound at the conclusion of the index procedure and assessed by an independent core laboratory

SECONDARY OUTCOMES:
Secondary safety endpoint: Absence of Major Adverse Events | 180 days, 12 months,vand 24 months post index procedure.
  Absence of Major Adverse Events (MAEs)
Secondary safety endpoint: Procedure related complications | 30 days, 6 months, 12 months, and 24 months post index procedure
  Procedure related complications
Secondary safety endpoint: Device related complications | 30 days, 6 months, 12 months, and 24 months post index procedure
  Device related complications. Device related complications are defined as device fracture(s), device migration, and device occlusion requiring intervention.
Secondary effectiveness endpoint: Freedom of aneurysmal sac enlargement | Day 30, 12 months, and 24 months post index procedure
  Freedom of aneurysmal sac enlargement. Enlargement is defined as a maximum diameter increase of > 5 mm per year, or aneurysm sac volume increase of > 10% per year, as assessed by CT scans and an independent core laboratory
Secondary effectiveness endpoint: Aneurysmal sac shrinkage | Day 30, 12 months, and 24 months post index procedure
  Aneurysmal sac shrinkage. Shrinkage is defined as a maximum diameter decrease of > 5 mm per year, or aneurysm sac volume decrease of > 10% per year, as assessed by CT scans and an independent core laboratory
Secondary effectiveness endpoint: Technical Success | Day 30
  Technical Success, defined as the presence of the device in the intended location and absence of device occlusion as assessed by CT scans and an independent core laboratory
Secondary effectiveness endpoint: Immobilization of the distal AAA neck | Day 30, 6 months, 12 months and 24 months
  Immobilization of the distal AAA neck, defined as aortic circumferential cyclic strain < 10% as measured via vascular ultrasound and assessed by an independent core laboratory
Secondary effectiveness endpoint: Absence of requirement of AAA repair | 30 days, 6 months, 12 months, and 24 months post index procedure.
  Absence of requirement of AAA repair (OR or EVAR)
Secondary effectiveness endpoint: Absence of aneurysm related mortality | 6 months, 12 months, and 24 months post index procedure
  Absence of aneurysm related mortality

OTHER OUTCOMES:
Quality of Life (QoL) | 6 months, 12 months, 4 months
  Short Form-36 (SF-36) Health Survey will be used to assess quality of life. The scale ranges from 0 to 100, where higher scores represent better quality of life. Subscale scores (each 0-100, higher is better) will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Raaz, MD, Study Director — Angiolutions GmbH
Locations (1):
- Еzgu Niyат Llc, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No